CLINICAL TRIAL: NCT04431830
Title: Meaning-Centered Pain Coping Skills Training: A Randomized Pilot Trial for Patients With Advanced Cancer and Pain
Brief Title: Meaning-Centered Pain Coping Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00105953
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumor; Pain
Keywords: Solid Tumor Cancer; Pain; Meaning-Centered Psychotherapy; Pain Coping Skills Training; Meaning-Centered Pain Coping; Advanced Cancer
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an intervention or a standard care control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning-Centered Pain Coping Skills Training (Experimental): Four, 45-60 minute, videoconference-delivered sessions focus on training participants in cognitive and behavioral skills (e.g., guided imagery) for managing pain.
  Interventions: Behavioral: Meaning-Centered Pain Coping Skills Training
- Standard Care (No Intervention): Information and referrals for free services available through the Duke Cancer Patient Support Program.

INTERVENTIONS:
Behavioral: Meaning-Centered Pain Coping Skills Training — The goal of this intervention is to help participants manage pain so that they can engage with what gives them a sense of meaning, purpose, and significance in life.
  Arms: Meaning-Centered Pain Coping Skills Training

SUMMARY:
This study is a randomized clinical trial of a psychosocial pain management intervention called, Meaning-Centered Pain Coping Skills Training (MCPC). Patients with advanced solid tumor cancer and at least moderate pain will be randomized to MCPC or a standard care control condition. Patient-reported outcomes will be assessed at baseline and 5- and 10-week follow-ups. The first aim of this study is to assess the feasibility of conducting a randomized clinical trial to test MCPC. The second aim is to characterize MCPC's effects on patient-reported outcomes of pain severity, pain interference, meaning in life, self-efficacy for pain management, and psychological distress. The third aim is to describe participants' experiences of MCPC using semi-structured qualitative interviews. The risk and safety issues in this trial are low and limited to those common to a psychosocial intervention (e.g., loss of confidentiality).

DETAILED DESCRIPTION:
Many patients with advanced cancer describe pain as their most feared and distressing symptom. In this population, higher pain levels often predict worse physical, emotional, and existential/spiritual well-being. Psychosocial interventions show promise for improving cancer-related pain; however, no interventions address existential concerns (e.g., a loss of meaning in life) that are common among those facing pain from advanced illness. To address this need, an intervention called Meaning-Centered Pain Coping Skills Training (MCPC) was developed. MCPC seeks to teach patients cognitive and behavioral skills for managing pain (e.g., guided imagery) in order to help them engage with what gives their life a sense of meaning, purpose, and significance.

This pilot study is being conducted to prepare for a large-scale clinical trial that will test the efficacy of MCPC for improving patients' pain and pain-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV solid tumor cancer diagnosis; or stage III pancreatic or lung cancer diagnosis
* At least moderate pain (worst pain in past week >/= 4 out of 10) at screening
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2 at screening
* Ability to speak and read English

Exclusion Criteria:

* Brain tumor diagnosis
* Significant cognitive impairment
* Untreated serious mental illness that would interfere with engagement in the interventions (e.g., schizophrenia)
* Previous engagement in Pain Coping Skills Training or Meaning-Centered Psychotherapy
* Enrollment in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual | Baseline
  Treatment feasibility will be evidenced by meeting study accrual (N = 60).
Feasibility as measured by adherence and assessment completion | 5-week follow-up (immediately post-intervention)
  Treatment feasibility will be evidenced by at least 75% of participants completing all four intervention sessions as well as the 5-week follow-up assessment.
Feasibility as measured by attrition | 5-week follow-up (immediately post-intervention)
  Treatment feasibility will be evidenced by no more than 25% attrition by the 5-week follow-up.

SECONDARY OUTCOMES:
Change in pain severity | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Pain severity will be measured using the Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF consists of 4 items assessing pain severity, including worst, least, average, and current pain. The minimum value on this scale is 0 and the maximum value is 10. Higher scores represent worse outcomes.
Change in pain interference | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Pain interference will be measured using the 6-item Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference-Short Form. This measure assesses the degree to which pain has impacted patients' enjoyment of life and engagement in social, cognitive, emotional, physical, and recreational activities. The minimum value on this scale is 6 and the maximum value is 30. Higher scores represent worse outcomes.
Change in meaning in life | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Meaning in life (i.e., purpose, coherence, and significance) and overall spiritual well-being will be measured using the 12-item Functional Assessment of Cancer Therapy - Spiritual Well-Being scale (FACIT-Sp).The minimum value on each subscale is 0 and the maximum value is 4. Higher scores represent better outcomes.
Change in self-efficacy for pain management | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Self-efficacy for pain management will be measured using the Self-efficacy for Pain Management subscale of the Chronic Pain Self-Efficacy Scale. The subscale includes 5 items assessing patients' confidence regarding pain management, managing pain during daily activities, keeping pain from interfering with sleep, and confidence in their ability to reduce pain using methods other than taking additional medication.The minimum value on this scale is 10 and the maximum value is 100. Higher scores represent better outcomes.
Change in anxiety | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Anxiety will be measured using the 7-item version of the Generalized Anxiety Disorders scale (GAD-7), which assesses the frequency of nervousness, worry, difficulty relaxing, restlessness, irritability, and fear. The minimum value on this scale is 0 and the maximum value is 21. Higher scores represent worse outcomes.
Change in depressive symptoms | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Depressive symptoms will be measured using the 8-item version of the Patient Health Questionnaire (PHQ-8), which assesses the frequency of anhedonia, depressed mood, sleep difficulties, lack of energy, appetite disturbance, low self-esteem, trouble concentrating, and psychomotor retardation.The minimum value on this scale is 0 and the maximum value is 24. Higher scores represent worse outcomes.
Change in hopelessness | Baseline, 5-week follow-up (immediately post-intervention), and 10-week follow-up
  Hopelessness will be measured using the Hopelessness Assessment in Illness Questionnaire. The scale includes 8 items assessing the degree to which patients have felt hopelessness, discouragement, and dread. The minimum value on this scale is 0 and the maximum value is 16. Higher scores represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Winger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winger JG, Kelleher SA, Ramos K, Check DK, Yu JA, Powell VD, Lerebours R, Olsen MK, Keefe FJ, Steinhauser KE, Porter LS, Breitbart WS, Somers TJ. Meaning-centered pain coping skills training for patients with metastatic cancer: Results of a randomized controlled pilot trial. Psychooncology. 2023 Jul;32(7):1096-1105. doi: 10.1002/pon.6151. Epub 2023 May 12. PMID 37173865